CLINICAL TRIAL: NCT02479958
Title: A Randomized in Vitro Evaluation of Antimicrobial Photodynamic Therapy on Deciduous Carious Dentin
Brief Title: An in Vitro Evaluation of Antimicrobial Photodynamic Therapy on Deciduous Carious Dentin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carolina Steiner-Oliveira, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150/10
Record Dates: First submitted 2015-05-25; First posted 2015-06-24 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Dental Caries
Keywords: Photochemotherapy; Bacteria
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental)
  Interventions: Procedure: Rubber dam isolation; Procedure: Tooth drying; Procedure: Dentin wash with chlorhexidine 2%
- APDT 1 (Experimental)
  Interventions: Procedure: Rubber dam isolation; Procedure: Tooth drying; Procedure: Antimicrobial Photodynamic Therapy 1
- APDT 2 (Experimental)
  Interventions: Procedure: Rubber dam isolation; Procedure: Tooth drying; Procedure: Antimicrobial Photodynamic Therapy 2

INTERVENTIONS:
Procedure: Rubber dam isolation — Tooth was isolated using a rubber dam isolation in order to collect the dentin samples
Procedure: Tooth drying — The tooth was dried with air jet.
Procedure: Dentin wash with chlorhexidine 2% — Partial carious tissue was removed with conventional dentinal curette and collection of dentin with a micropunch (Ø = 1mm) was performed. The remaining dentin was washed with chlorhexidine 2%. After that a a new dentin collection was performed at another site of the cavity, and restoration with resin-modified glass ionomer cement was placed.
  Arms: Control
Procedure: Antimicrobial Photodynamic Therapy 1 — Partial carious tissue was removed with conventional dentine curette and collection of dentin with a micropunch (Ø = 1mm) was performed. The remaining dentin was washed with 200 µL of O-Toluidine blue dye (0.1 mg/mL) for 60 s. After this, a red LED light source with wavelength of 630 nm was used at 100 mW power, 9.0 J of energy, for 60 s with energy density of 30.0 J/cm2 . A new dentin collection was performed after this treatment at another site of the cavity and restoration with resin-modified glass ionomer cement Vitremer was placed.
  Arms: APDT 1
Procedure: Antimicrobial Photodynamic Therapy 2 — Partial carious tissue was removed with conventional dentine curette and initial collection of dentin with a micropunch (Ø = 1mm) was performed. Treatment of the remaining dentin was performed with 200 µL of methylene blue dye 0.01% for 5 min and after this, a red low level LASER light source with wavelength of 660 nm was used at 100 mW power, 9.0 J of energy, for 90 s with energy density of 320.0 J/cm2 . A new dentin collection was performed after this treatment at another site of the cavity and restoration with resin-modified glass ionomer cement was placed.
  Arms: APDT 2

SUMMARY:
Despite of the decline of dental caries, this disease is still common in polarized groups affecting children. Therefore, the aim of this randomized blind in vivo study was to compare the antimicrobial effect of two antimicrobial therapies in deciduous carious dentin. Thirty two patients aging from 5 to 7 years old had partial caries removal in deep carious dentin lesion in deciduous molar and were divided in three groups: 1. Control - chlorhexidine and resin modified glass ionomer cement (RMGIC); 2. LEDTB - antimicrobial photodynamic therapy (APDT) with LED (light emission diode) associated with toluidine blue orto dye solution and RMGIC; 3. LMB - APDT with laser associated with methylene blue dye solution and RMGIC. The patients were submitted to initial clinical and radiographic examination and demographic features were evaluated by biofilm, gingival, and dmft/dmfs indexes, besides clinical and radiographic follow up at 6 and 12 months after the treatments. The carious dentin was collected before and after each treatment and the number of Streptococcus mutans, Streptococcus sobrinus, Lactobacillus casei, Fusobacterium nucleatum, Atopobium rimae and total bacteria were established by quantitative PCR.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria consisted of good general health, without syndromes or chronic systemic diseases. They should also have at least one primary molar with deep carious lesion (2/3 of dentin) without pain symptomatology and compatible with reversible pulpits.

Exclusion Criteria:

* Children whose parents refused to sign the informed consent document, who did not cooperate with the clinical exams, whose teeth had the treatment choice changed (pain or evolution to irreversible pulpits), who did not attend to the appointments for the scheduled treatments, or who needed antibiotics treatment for other medical reasons were excluded from the study without prejudice.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quantification of Bacteria by quantitative Polymerase Chain Reaction (PCR) | 15 days after dentin collection
  Quantification of S. mutans, L. casei, F. nucleatum, A. rimae and total bacteria by PCR (Polymerase Chain Reaction)

SECONDARY OUTCOMES:
Tooth Pain | 6 months
  Patients reported the presence or absence of tooth pain after 6 months
Tooth Pain | 12 months
  Patients reported the presence or absence of tooth pain after 6 months
Restoration Quality | 6 months
  The quality of restoration was evaluated through the absence of radiographic radiolucent area after 6 months
Restoration Quality | 12 months
  The quality of restoration was evaluated through the absence of radiographic radiolucent area after 12 months